CLINICAL TRIAL: NCT02627534
Title: Local Effects of Adjunct Photodynamic Therapy in the Treatment of Type 2 Diabetic Patients With Chronic Periodontitis: Split-mouth Randomized Triple-blind Clinical Trial
Brief Title: Effects of Adjunct Photodynamic Therapy in the Treatment of Type 2 Diabetic Patients With Chronic Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Nídia Cristina Castro dos Santos, DDS, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NSFOSJC
Record Dates: First submitted 2015-11-25; First posted 2015-12-11 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Periodontitis; Diabetes Mellitus
Keywords: Photodynamic therapy; Ultrasonic debridement; Chronic periodontitis; Type 2 diabetes
MeSH Terms: conditions — Chronic Periodontitis; Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasonic Debridement (UD) (Active Comparator): Ultrasonic Debridement (UD) (n=20)
  Interventions: Procedure: Ultrasonic debridement
- UD + Antimicrobial Photodynamic Therapy (Experimental): Ultrasonic Debridement + aPDT (UD+aPDT) (n=20)
  Interventions: Procedure: Ultrasonic debridement; Procedure: Antimicrobial photodynamic therapy

INTERVENTIONS:
Procedure: Ultrasonic debridement — All periodontal pockets received ultrasonic debridement (Cavitron, Dentsply) with specific inserts (UI25KSF10S, Hu-Friedy). All diseased sites were instrumented in one session by an experienced periodontist.
Procedure: Antimicrobial photodynamic therapy — After ultrasonic debridement, one randomly selected periodontal pocket received an additional aPDT performed by a trained operator (NMRBA). One pocket with probing depth ≥ 5mm in each patient was randomly selected to aPDT. After washing the pocket with saline solution, the photosensitizer (methylene blue 10mg/ml) was applied to the bottom of the pocket in a coronal direction. Following this, the pocket was exposed to a diode laser light with a fibre optic application for 1 min (Thera Lase DMC - Brazil), with wavelength of 660nm, power of 60mW and fluency of 129J/cm2.
  Arms: UD + Antimicrobial Photodynamic Therapy

SUMMARY:
Periodontal Diseases are considered the sixth complication of Diabetes Mellitus (DM). This close relationship between both diseases is characterized by mutual influence. The presence of DM might impair prognosis of diverse dental treatments due to its inflammatory nature, negative influence on wound healing, on bone biology, and the establishment of infections. Consequently, knowledge of new dental therapies and the biology of dental treatments for chronic periodontitis in diabetic patients can enhance quality of life and make these treatments more adequate for this common profile of patients.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) has become a global epidemic. Its complications can have a significant impact on quality of life, longevity, and costs in public health. The World Health Organization (WHO) estimates that by 2030, 439 million people will suffer from diabetes, around 10% of the world adult population (WHO, 2011). Periodontal Diseases are considered the sixth complication of DM. This close relationship between both diseases is characterized by mutual influence. Thus, an appropriate control of periodontal disease may facilitate the DM control, improving quality of life on diabetes patients. Besides that, the presence of DM might impair prognosis of diverse dental treatments due to its inflammatory nature, negative influence on wound healing, on bone biology, and the establishment of infections. Consequently, knowledge of new dental therapies and the biology of dental treatments for chronic periodontitis in diabetic patients can enhance quality of life and make these treatments more adequate for this common profile of patients. Therefore, the aim of the present study is to investigate the effectiveness of antimicrobial photodynamic therapy as adjunct to full-mouth debridement for the treatment of periodontitis in type 2 diabetic patients through a split-mouth randomized triple-blind clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of type 2 DM for ≥5 years
* DM treatment with oral hypoglycemic agents or insulin supplementation and diet
* glycated hemoglobin (HbA1c) levels from 6.5% to 11%
* at least 15 teeth (excluding third molars and teeth indicated for extraction)
* moderate to severe generalized chronic periodontitis (Armitage, 1999)
* agree and sign the formal consent to participate in the study after receiving an explanation of risks and benefits from an individual who was not a member of the study (Resolution number 196 - October, 1996, and Ethics and Code of Professional Conduct in Dentistry - CFO179/93).

Exclusion Criteria:

* medical conditions that required prophylactic antimicrobial coverage
* SRP in the previous 6 months
* antimicrobial therapies in the previous 6 months
* anti-inflammatory therapies in the previous 6 months
* systemic conditions, other than DM, that could affect the progression of chronic periodontitis
* current use of medication that could interfere with periodontal response to treatment
* pregnancy or lactation
* smoking

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2015-03 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Probing Depth | Reductions in Probing Depth was compared at baseline and 180 days
  Assessed with manual probe (North Carolina, Hu-Friedy)

SECONDARY OUTCOMES:
Clinical Attachment Level | Clinical Attachment Level gain was compared at baseline and 180 days
  Assessed with manual probe (North Carolina, Hu-Friedy)

OTHER OUTCOMES:
Gingival Recession | Gingival Recession changes was compared at baseline and 180 days
  Assessed with manual probe (North Carolina, Hu-Friedy)

CONTACTS AND LOCATIONS:
Overall Officials: Mauro P Santamaria, PhD, Study Director — ICT - UNESP
Locations (1):
- Instituto de Ciência e Tecnologia de São José dos Campos - UNESP, Sâo José Dos Campos, São Paulo, Brazil

REFERENCES:
- [Derived] Castro Dos Santos NC, Andere NM, Araujo CF, de Marco AC, Dos Santos LM, Jardini MA, Santamaria MP. Local adjunct effect of antimicrobial photodynamic therapy for the treatment of chronic periodontitis in type 2 diabetics: split-mouth double-blind randomized controlled clinical trial. Lasers Med Sci. 2016 Nov;31(8):1633-1640. doi: 10.1007/s10103-016-2030-8. Epub 2016 Jul 22. PMID 27448223